CLINICAL TRIAL: NCT02618473
Title: Impact of a Motion Correction Algorithm on Image Quality and Diagnostic Utility in Patients Undergoing CT Angiography: A Randomized Controlled Trial
Brief Title: Effect of Snapshot Freeze on Cardiac CT Image Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Hussam Mahmoud Sheta, M.D, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Snapshot Freeze
Record Dates: First submitted 2015-11-18; First posted 2015-12-01 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-11

CONDITIONS: Heart Diseases
Keywords: Coronary computed tomography angiography; motion artifacts; motion correction algorithm; diagnostic utility
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- seloken (No Intervention): In "seloken" arm, patients performs the cardiac CT procedure regarding the national scan guidelines, ande receive 5-10 intravenous seloken, until heart rate below 60 beats pr minit is achieved.
- non-seloken (Experimental): Patients randomized to "non-seloken", do not receive any medication.
  Interventions: Other: non-seloken

INTERVENTIONS:
Other: non-seloken — regarding the guidelines patients receive seloken before the cardiac CT scan to lower the heart rate during the scan. The intervention in this study is to avoid the medication with seloken before the scan, and to investigate if the use of a new motion correction scan algorithm can compensate for the absence of the seloken.
  Arms: non-seloken

SUMMARY:
The aim of this study was to investigate the effect of a new motion correction algorithm on image quality and diagnostic utility in unselected patients undergoing coronary cardiac computed tomography, and to investigate if this motion correction algorithm can compensate for the usual use of intravenously medication (beta-blockers) before the scan.

DETAILED DESCRIPTION:
Aims:

To investigate the motion correction algorithm Snapshot-Freeze(SSF) compared to standard reconstruction(STD) in patients randomized to receive beta-blockers(BB) or no beta-blockers(non-BB) before coronary CT angiography (CCTA), and to investigate if SSF can replace BB.

Methods:

The study included 140 consecutively recruited patients scheduled to CCTA to rule out coronary artery disease.

The inclusion criteria were: age ≥ 18 years, Glomerular filtration rate ≥ 60 mL/min, Heart Rate between 60 and 85 bpm before the scan. The exclusion criteria were: irregular heart rhythm or history of allergic reaction to contrast agents. Patients were randomized to the BB group or the non-BB group. The trial complied with the Declaration of Helsinki and was approved by the local ethics committee. Written informed consent was obtained from all patients.

Image quality score:

The evaluation was performed according to the Likert score as follows: 1: excellent, no motion artifacts, clear delineation of the segments; 2: good, minor artifacts, mild blurring of the segment; 3: adequate, moderate artifacts, moderate blurring without structure discontinuity; and 4: poor and non-diagnostic, with doubling or discontinuity in the course of the segments, preventing evaluation or producing vessel structures that were not differentiable. In cases where the image quality was less than excellent (Likert score 2-4), the readers noted the reason(s) for the observed artifact.

Statistical analyses:

Quantitative variables were expressed as mean ± standard deviation, and categorical values as frequencies or percentages. Values from the Likert score were dichotomized to excellent vs. non-excellent (Likert score 1 vs. 2-4), and diagnostic vs. non-diagnostic (Likert score 1-3 vs. 4). McNemar's test was performed to test categorical variables separately per-vessel and per-patient level. Analyses for all segments were calculated by the Wilcoxon signed-rank test.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years,
* glomerular filtration rate ≥ 60 mL/min,
* heart rate between 60 and 85 bpm before the scan

Exclusion Criteria:

* irregular heart rhythm
* history of allergic reaction to contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
images with non diagnostic image quality | up to 1 year
  number of non diagnostic images.

SECONDARY OUTCOMES:
images with Excellent image quality | up to 1 year
  number of presented images with "Excellent" image quality
motion artifacts | up to 1 year
  number of presented motion artifacts

CONTACTS AND LOCATIONS:
Overall Officials: jess Lambrechtsen, MD, Study Director — Odense University Hospital
Locations (1):
- Department of Medical Research, OUH, Svendborg, Svendborg, Svendborg, Denmark